CLINICAL TRIAL: NCT01855802
Title: Greek Physicians Perceptions Regarding Generics Prescribing in Glaucoma
Status: Completed | Type: Observational
Sponsor: Democritus University of Thrace (Other)
Responsible Party: Principal Investigator, Georgios Labiris, Assistant Professor, Democritus University of Thrace
Other Study IDs: EIT-GG-P
Record Dates: First submitted 2013-04-30; First posted 2013-05-17 (Estimated); Last update posted 2017-01-18 (Estimated); Status verified 2017-01

CONDITIONS: Glaucoma
Keywords: Greece; Ophthalmology; Glaucoma; Generics; Perception
MeSH Terms: conditions — Glaucoma

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

SUMMARY:
This attempts to investigate the perceptions of Greek Ophthalmologists regarding generics prescription in glaucoma by means of a structured questionnaire.

DETAILED DESCRIPTION:
The following dimensions will be recorded

1. Overall physician's empathy regarding generics in glaucoma
2. Physician's prescribing habits regarding generics in glaucoma
3. Physician's perceptions regarding generics cost-effectiveness in glaucoma
4. Physician's perceptions regarding adequacy of Greek regulatory authorities (generic market in glaucoma)
5. Physician's perceptions regarding adequacy of European regulatory authorities (generic market in glaucoma)

ELIGIBILITY:
Inclusion Criteria:

Licensed Registration to Greek Ophthalmology Council

Exclusion Criteria:

-

Ages: 25 Years to 67 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Greek Medical Council Members
Sampling Method: Non-Probability Sample
Enrollment: 70 (Actual)
Dates: Start 2013-04; Primary Completion 2013-09 (Actual); Study Completion 2013-10 (Actual)

PRIMARY OUTCOMES:
Generic Perception | 3 months

CONTACTS AND LOCATIONS:
Overall Officials: Georgios Labiris, PhD, Principal Investigator — Democritus University of Thrace, Medical School
Locations (1):
- University Hospital of Alexandroupolis, Alexandroupoli, Evros, Greece

REFERENCES:
- [Result] Labiris G, Fanariotis M, Kastanioti C, Alexias G, Protopapas A, Karampitsakos T, Niakas D. Greek Physicians' Perceptions on Generic Drugs in the Era of Austerity. Scientifica (Cairo). 2015;2015:251792. doi: 10.1155/2015/251792. Epub 2015 Sep 17. PMID 26457225